CLINICAL TRIAL: NCT06203509
Title: An Equity-focused Intervention to Improve Care Transitions for Medicaid Insured Individuals With Co-occurring Chronic Medical Conditions and Serious Mental Illness
Brief Title: Improving Care Transitions for Medicaid Insured Individuals With Co-occurring Serious Mental Illness
Acronym: THRIVE-SMI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R18HS029815-01 (AHRQ); 1R18HS029815-01 (AHRQ)
Record Dates: First submitted 2024-01-02; First posted 2024-01-12 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Care Transitions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- THRIVE Intervention (Experimental): THRIVE Intervention
  1-month intensive post discharge case management and care coordination
  Interventions: Behavioral: Thrive Intervention
- Usual Care (No Intervention): Discharge to home without intensive post-acute case management or care coordination.

INTERVENTIONS:
Behavioral: Thrive Intervention — • The THRIVE Clinical Pathway is a standardized transitional care clinical pathway that supports Medicaid insured or Medicaid eligible individuals being managed for both chronic diseases and serious mental illness following hospitalization.
  Arms: THRIVE Intervention

SUMMARY:
This study aims to evaluate the THRIVE clinical pathway at HUP, focusing on supporting Medicaid-insured individuals, including those with serious mental illness, following hospitalization. The study will assess clinician/administrator perspectives on the pathway's feasibility, appropriateness, and acceptability and analyze referral patterns and post-discharge outcomes.

The objectives are:

1. To conduct a qualitative study evaluating the implementation of THRIVE, particularly its adaptation to include patients with serious mental illness.
2. To examine referral patterns, 30-day readmission rates, and ED utilization for THRIVE participants, comparing them with those receiving standard care.

Participants will be referred to home care services during hospitalization and seen by a home care nurse within 48 hours post-discharge. A discharging physician or Advanced Practice Provider will oversee care for 30 days or until a primary care or specialist visit. The Care Coordination Team will hold weekly case conferences for 30 days post-discharge to address both health and mental health needs. The study will compare outcomes of Medicaid-insured patients, including those with serious mental illness, to those receiving usual care.

DETAILED DESCRIPTION:
Detailed Description:

This study is a single-site Type 1 hybrid effectiveness-implementation parallel mixed methods (quantitative + qualitative) quasi-experimental study at HUP, focusing on the THRIVE clinical pathway. It integrates simultaneous quantitative and qualitative data collection and analysis, with a stronger emphasis on quantitative data to evaluate referrals, outcomes, and program fidelity. The qualitative aspect will explore the implementation process, delving into the barriers and facilitators encountered by healthcare providers. It will also assess stakeholder perspectives on the intervention's impact on health inequities among Medicaid-insured individuals in both acute and home care settings. By nesting qualitative interviews within a quasi-experimental framework, the study aims to examine the intervention's effect on primary outcomes (homecare referrals, 30-day readmission, ED utilization, connection to PCP) and to identify professional and organizational barriers to its implementation. The combination of effectiveness data with contextual insights will inform understanding of factors critical to THRIVE's implementation and outcomes.

Qualitative Study:

The recruitment process is meticulously managed to track each participant's journey. Recruitment begins in early January, with participants contacted via email, providing study details and interview scheduling links. Follow-up reminders ensure participant engagement. Interviews, conducted virtually and recorded with consent, focus on maintaining confidentiality and privacy. Non-consented sessions are captured through detailed notes. Post-interview, recordings are transcribed for analysis, enabling categorization into codes and themes for a deeper understanding of participant perspectives.

Quantitative Study:

Employing a stepped wedge design, the study would begin early March and would involve a randomized training of case managers at HUP over several months. Initially, a subset of case managers receives training on the THRIVE pathway and starts offering referrals. After 8 weeks, the remaining case managers are trained and begin making referrals. This staggered approach allows for evaluation of the THRIVE intervention's rollout and its impact on patient care and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Medicaid insured
* Residing in the state of Pennsylvania
* Experienced a hospitalization at study hospital
* Agrees to home care at partner home care setting.

Exclusion Criteria:

* Individuals under age 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 267 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Rates of Referrals to Homecare | Through study completion, an average of 18 months
  We will evaluate changes in home care referrals between case managers exposed to the intervention compared to those who were not
Rates of Readmissions | 30 days following hospital discharge
  We will evaluate the rate of readmissions over the course of the study for THRIVE participants compared to those receiving usual care
Rates of Emergency Department Visit | 30 days following hospital discharge
  We will evaluate the rate of ED visits over the course of the study for THRIVE participants compared to those receiving usual care.
Primary Care or Specialist Visit | 30 Days following hospital discharge
  We will compare the rates of primary care provider and specialist visits within 30 days following discharge compared to those receiving usual care

SECONDARY OUTCOMES:
Feasibility, Acceptability, Appropriateness, Workload | Through study completion, an average of 18 months
  We will conduct interviews of clinicians at the conclusion of the study to gather perceptions of the THRIVE clinical pathway and facilitators and barriers to engaging with the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline M Brooks Carthon, PhD,RN, Principal Investigator — University of Pennsylvania
Locations (1):
- Upenn School of Nursing Centre For Health Outcomes Policy Research, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brooks Carthon JM, Tibbitt C, Amenyedor KE, Bettencourt AP, Babe E, Cacchione PZ, Brom H. Pre-Implementation Strategies to Support Adaptation of Thrive: A Care Transitions Model for Economically Disadvantaged Patients with Serious Mental Illness. Nurs Rep. 2024 Dec 2;14(4):3803-3818. doi: 10.3390/nursrep14040278. PMID 39728639
- [Derived] Brooks Carthon JM, Brom H, Amenyedor KE, Harhay MO, Grantham-Murillo M, Nikpour J, Lasater KB, Golinelli D, Cacchione PZ, Bettencourt AP. Transitional Care Support for Medicaid-Insured Patients With Serious Mental Illness: Protocol for a Type I Hybrid Effectiveness-Implementation Stepped-Wedge Cluster Randomized Controlled Trial. JMIR Res Protoc. 2024 Nov 12;13:e64575. doi: 10.2196/64575. PMID 39531274